CLINICAL TRIAL: NCT02178605
Title: A Prospective Non-Randomized Investigation Of The Use Of Infuse® (rhBMP-2) In Cervical Arthrodesis
Brief Title: rhBMP-2 in Cervical Arthrodesis
Status: Completed | Type: Observational
Sponsor: Virginia Spine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 08-07
Record Dates: First submitted 2014-06-26; First posted 2014-07-01 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2016-10

CONDITIONS: Cervical Arthrodesis
Keywords: rhBMP-2; arthrodesis; cervical
MeSH Terms: conditions — Ankylosis | interventions — Bone Morphogenetic Protein 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical arthrodesis candidates: Patients scheduled to undergo cervical arthrodesis to treat their spinal pathology will undergo cervical arthrodesis with rhBMP-2
  Interventions: Procedure: Cervical arthrodesis with rhBMP-2

INTERVENTIONS:
Procedure: Cervical arthrodesis with rhBMP-2 — Cervical arthrodesis with rhBMP-2
  Other Names: Infuse

SUMMARY:
This prospective study will investigate the use of recombinant human bone morphogenetic protein (rhBMP-2) in the current surgical standard of care for cervical spine pathology. Specifically, the outcomes of three forms of cervical fusion will be investigated:

1. Anterior cervical fusion with rhBMP-2, allograft corticocancellous bone as an interbody device, and anterior cervical plate fixation.
2. Posterior cervical fusion with rhBMP-2, local bone graft, with or without posterior screw fixation.
3. A combination of the previous two approaches: a combined anterior-posterior cervical fusion with rhBMP-2.

DETAILED DESCRIPTION:
SURGICAL TECHNIQUES

1. Anterior cervical fusion The technique of anterior cervical discectomy and arthrodesis of the spine has been previously described by Smith-Robinson (ref) and is an accepted technique for anterior cervical fusion. Upon completion of adequate decompression, a gentle distraction maneuver may be performed by using either Caspar distraction pins or an interbody spreading device, taking care to avoid injury to the endplates.

   The endplates are then prepared with the use of a rasp or high speed burr taken to both superior and inferior endplates to remove the cartilagenous material and identify the bony endplate. Once hemostasis is obtained, the appropriate size allograft implant is chosen. That implant is then defrosted and brought into the surgical field. Concurrently, rhBMP-2 ((INFUSE®) Medtronic, Inc. Minneapolis, MN) has been reconstituted with sterile water, placed on an absorbable (type I bovine) collage sponge (ACS), cut to deliver the appropriate dose to each spinal level and is on the field as well. The partial BMP/ACS sponge is inserted into each disc space level, posterior to the structural implant. The dosage of rhBMP-2 used is approximately 0.525 mg per disc level or interbody space treated.

   The interbody device utilized is LifeNet Health's VertiGraft® VG2®. In the case of these allograft intervertebral implants, product safety and efficacy has been validated and patented by LifeNet Health using both an Allowash® and Allowash XG® technology. This is an intensive decontamination, disinfection and scrubbing regimen to remove and inactivate both viruses and bacteria which may be present from the donor harvesting process. The Allowash® process removes virtually all cellular elements of the bone thereby providing an additional line of defense against infectious disease. The second step consists of terminal sterilization of the cortico-cancellous allograft tissue. These processes have been validated and render the tissue sterile without compromising either the biomechanical or biochemical properties of allograft tissue intended for spinal applications.

   Plate fixation with the Atlantis® Cervical Plate (Medtronic, Inc. Minneapolis, MN) is carried out by serially drilling each of the screw holes and placing the appropriate length (3.5 x 14-15 mm) screw into each of the holes. The locking screw mechanism on the plate is then secured and a lateral cervical radiograph is called for to confirm appropriate levels and instrumentation placement. A medium Hemovac drain is placed in the anterior prevertebral space and brought out through a separate stab incision. Routine closure is then carried out.
2. Posterior Cervical Arthrodesis A longitudinal incision is made in the midline of the posterior neck, directly over the involved spinal level(s). The fascia and muscle are gently divided, exposing the spinous processes and lamina. An x-ray is obtained to confirm the appropriate spinal levels to be fused. A laminectomy and foraminotomy can be performed if necessary. Two (3.5 mm x 14mm) cortical screws ((Vertex (TM) Medtronic, Inc. Minneapolis, MN) are affixed to each lateral mass in the method previous described by Magerl (ref) and connected with a titanium rod on each side of the spine. The bony surfaces and facet joints are then decorticated. One sponge of the BMP/ACS product is placed over the decorticated bone surfaces on each side. The bone removed during the decompresion laminectomy is morsellized and placed in and around the facet joints. The amount of rh-BMP-2 used will be a total of 2.1 mg placed bilaterally, to a total of 4.2mg.
3. Combined Anterior-Posterior Cervical Arthrodesis This surgical procedure combines a posterior cervical decompression and fusion with an anterior cervical fusion. The techniques described for the individual surgical procedures are applicable to the combined Anterior-Posterior procedure. In an anterior-posterior surgery, the amount and positioning of rhBMP-2 will be similar to the anterior surgery (0.525 mg placed anteriorly at each level) or similar to the posterior surgery (2.4 mg across the entire lateral mass on each side posteriorly).

ELIGIBILITY:
Inclusion Criteria:

* Has cervical spine pathology as noted by neck pain with or without arm symptoms, functional deficit and/or neurological deficit, confirmed by patient history, as well as radiographic imaging studies:

  * CT, MRI scan, x-ray imaging are to include one or more of the following:
  * Instability, as defined by translational motion greater than or equal to 3.5 mm or angular motion greater than 11° at a single segment based upon flexion/extension radiographs.
  * Osteophyte formation.
  * Decreased disc space height.
  * Facet joint degeneration.
  * Disc herniation or protrusion.
  * Signs or symptoms of spinal cord compression (i.e., myelopathy).
* One or more symptomatic levels of degeneration between C3 and C7.
* Age 18 years of age or older at the time of surgery.
* Has not responded to nonoperative treatments including restricted activity, physical therapy, medications, corticosteroid injections, manipulation, TENS for a period of at least three months.
* If female of childbearing age who is not pregnant or nursing and who agrees to use adequate contraception for at least six months following surgery.
* Is willing and able to comply with the study protocol, sign the patient informed consent form, and able to sign the authorization to disclose health information consent form.

Exclusion Criteria:

* Has a condition which requires postoperative medications that interfere with fusion, such as steroids.
* Has been previously diagnosed with osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated.
* Has active malignancy.
* Has overt or active bacterial infection, either local or systemic.
* Has fever (temperature greater than 101° Fahrenheit oral at the time of surgery).
* Has a documented titanium alloy allergy or allergy to bovine collagen.
* Is mentally incompetent.
* Has a Waddell sign of inorganic behavior score of 3 or greater.
* Is a prisoner.
* Is an alcohol and/or drug abuser, as defined by currently undergoing treatment for alcohol and/or drug abuse.
* Has a history of autoimmune disease.
* Has a hypersensitivity to protein pharmaceuticals, monoclonal antibodies, gammaglobulin, or collagen.
* Has a history of endocrine of metabolic disorder known to affect osteogenesis.
* Is currently pregnant or plans on becoming pregnant within the six months following the surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at a single site and candidates for cervical arthrodesis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | Up to 2 years
  Number of Participants with Serious and Non-Serious Adverse Events intra-operative and up to 2 years post-operative

SECONDARY OUTCOMES:
Improvement in patient-reported outcomes | Pre-operative up to 2 years post-operative
  Change from pre-operative to 2-year post-operative n disability, neck pain, arm pain, and health

CONTACTS AND LOCATIONS:
Overall Officials: Brian R Subach, MD, Principal Investigator — Virginia Spine Institute
Locations (1):
- Virginia Spine Institute, Reston, Virginia, United States

REFERENCES:
- [Background] Ong KL, Villarraga ML, Lau E, Carreon LY, Kurtz SM, Glassman SD. Off-label use of bone morphogenetic proteins in the United States using administrative data. Spine (Phila Pa 1976). 2010 Sep 1;35(19):1794-800. doi: 10.1097/BRS.0b013e3181ecf6e4. PMID 20700081
- [Background] Perri B, Cooper M, Lauryssen C, Anand N. Adverse swelling associated with use of rh-BMP-2 in anterior cervical discectomy and fusion: a case study. Spine J. 2007 Mar-Apr;7(2):235-9. doi: 10.1016/j.spinee.2006.04.010. Epub 2006 Nov 20. PMID 17321975
- [Background] Mroz TE, Wang JC, Hashimoto R, Norvell DC. Complications related to osteobiologics use in spine surgery: a systematic review. Spine (Phila Pa 1976). 2010 Apr 20;35(9 Suppl):S86-104. doi: 10.1097/BRS.0b013e3181d81ef2. PMID 20407355
- [Background] Cahill KS, Chi JH, Day A, Claus EB. Prevalence, complications, and hospital charges associated with use of bone-morphogenetic proteins in spinal fusion procedures. JAMA. 2009 Jul 1;302(1):58-66. doi: 10.1001/jama.2009.956. PMID 19567440
- [Background] Williams BJ, Smith JS, Fu KM, Hamilton DK, Polly DW Jr, Ames CP, Berven SH, Perra JH, Knapp DR Jr, McCarthy RE, Shaffrey CI; Scoliosis Research Society Morbidity and Mortality Committee. Does bone morphogenetic protein increase the incidence of perioperative complications in spinal fusion? A comparison of 55,862 cases of spinal fusion with and without bone morphogenetic protein. Spine (Phila Pa 1976). 2011 Sep 15;36(20):1685-91. doi: 10.1097/BRS.0b013e318216d825. PMID 21897187
- [Background] Fineberg SJ, Ahmadinia K, Oglesby M, Patel AA, Singh K. Hospital outcomes and complications of anterior and posterior cervical fusion with bone morphogenetic protein. Spine (Phila Pa 1976). 2013 Jul 1;38(15):1304-9. doi: 10.1097/BRS.0b013e31828f494c. PMID 23462577
- [Background] Tumialan LM, Pan J, Rodts GE, Mummaneni PV. The safety and efficacy of anterior cervical discectomy and fusion with polyetheretherketone spacer and recombinant human bone morphogenetic protein-2: a review of 200 patients. J Neurosurg Spine. 2008 Jun;8(6):529-35. doi: 10.3171/SPI/2008/8/6/529. PMID 18518673
- [Background] Frenkel MB, Cahill KS, Javahary RJ, Zacur G, Green BA, Levi AD. Fusion rates in multilevel, instrumented anterior cervical fusion for degenerative disease with and without the use of bone morphogenetic protein. J Neurosurg Spine. 2013 Mar;18(3):269-73. doi: 10.3171/2012.12.SPINE12607. Epub 2013 Jan 25. PMID 23350532
- [Background] Lanman TH, Hopkins TJ. Early findings in a pilot study of anterior cervical interbody fusion in which recombinant human bone morphogenetic protein-2 was used with poly(L-lactide-co-D,L-lactide) bioabsorbable implants. Neurosurg Focus. 2004 Mar 15;16(3):E6. PMID 15198494
- [Background] Shields LB, Raque GH, Glassman SD, Campbell M, Vitaz T, Harpring J, Shields CB. Adverse effects associated with high-dose recombinant human bone morphogenetic protein-2 use in anterior cervical spine fusion. Spine (Phila Pa 1976). 2006 Mar 1;31(5):542-7. doi: 10.1097/01.brs.0000201424.27509.72. PMID 16508549
- [Background] Boakye M, Mummaneni PV, Garrett M, Rodts G, Haid R. Anterior cervical discectomy and fusion involving a polyetheretherketone spacer and bone morphogenetic protein. J Neurosurg Spine. 2005 May;2(5):521-5. doi: 10.3171/spi.2005.2.5.0521. PMID 15945426
- [Background] Stachniak JB, Diebner JD, Brunk ES, Speed SM. Analysis of prevertebral soft-tissue swelling and dysphagia in multilevel anterior cervical discectomy and fusion with recombinant human bone morphogenetic protein-2 in patients at risk for pseudarthrosis. J Neurosurg Spine. 2011 Feb;14(2):244-9. doi: 10.3171/2010.9.SPINE09828. Epub 2010 Dec 24. PMID 21184639
- [Background] Baskin DS, Ryan P, Sonntag V, Westmark R, Widmayer MA. A prospective, randomized, controlled cervical fusion study using recombinant human bone morphogenetic protein-2 with the CORNERSTONE-SR allograft ring and the ATLANTIS anterior cervical plate. Spine (Phila Pa 1976). 2003 Jun 15;28(12):1219-24; discussion 1225. doi: 10.1097/01.BRS.0000065486.22141.CA. PMID 12811263
- [Background] Smucker JD, Rhee JM, Singh K, Yoon ST, Heller JG. Increased swelling complications associated with off-label usage of rhBMP-2 in the anterior cervical spine. Spine (Phila Pa 1976). 2006 Nov 15;31(24):2813-9. doi: 10.1097/01.brs.0000245863.52371.c2. PMID 17108835
- [Background] Vaidya R, Carp J, Sethi A, Bartol S, Craig J, Les CM. Complications of anterior cervical discectomy and fusion using recombinant human bone morphogenetic protein-2. Eur Spine J. 2007 Aug;16(8):1257-65. doi: 10.1007/s00586-007-0351-9. Epub 2007 Mar 27. PMID 17387522
- [Background] Buttermann GR. Prospective nonrandomized comparison of an allograft with bone morphogenic protein versus an iliac-crest autograft in anterior cervical discectomy and fusion. Spine J. 2008 May-Jun;8(3):426-35. doi: 10.1016/j.spinee.2006.12.006. Epub 2007 Mar 7. PMID 17977799
- [Background] Lu DC, Tumialan LM, Chou D. Multilevel anterior cervical discectomy and fusion with and without rhBMP-2: a comparison of dysphagia rates and outcomes in 150 patients. J Neurosurg Spine. 2013 Jan;18(1):43-9. doi: 10.3171/2012.10.SPINE10231. Epub 2012 Nov 16. PMID 23157278
- [Background] Crawford CH 3rd, Carreon LY, McGinnis MD, Campbell MJ, Glassman SD. Perioperative complications of recombinant human bone morphogenetic protein-2 on an absorbable collagen sponge versus iliac crest bone graft for posterior cervical arthrodesis. Spine (Phila Pa 1976). 2009 Jun 1;34(13):1390-4. doi: 10.1097/BRS.0b013e3181a2da08. PMID 19440166
- [Background] Cimic M, Smoljanovic T, Bojanic I. Re: Hiremath GK, Steinmetz MP, Krishnaney AA. Is it safe to use recombinant human bone morphogenetic protein in posterior cervical fusion? Spine 2009;34:885-9. Spine (Phila Pa 1976). 2010 Feb 1;35(3):361; author reply 361-2. doi: 10.1097/BRS.0b013e3181cb4651. No abstract available. PMID 20118766
- [Background] Xu R, Bydon M, Sciubba DM, Witham TF, Wolinsky JP, Gokaslan ZL, Bydon A. Safety and efficacy of rhBMP2 in posterior cervical spinal fusion for subaxial degenerative spine disease: Analysis of outcomes in 204 patients. Surg Neurol Int. 2011;2:109. doi: 10.4103/2152-7806.83726. Epub 2011 Aug 13. PMID 21886882
- [Background] Hodges SD, Eck JC, Newton D. Retrospective study of posterior cervical fusions with rhBMP-2. Orthopedics. 2012 Jun;35(6):e895-8. doi: 10.3928/01477447-20120525-30. PMID 22691663
- See also: Virginia Spine Institute — http://www.spinemd.com/